CLINICAL TRIAL: NCT03441594
Title: Psychological Mechanisms Linking Food Insecurity and Obesity (Food Mind Pilot Study)
Brief Title: Psychological Mechanisms Linking Food Insecurity and Obesity
Status: Completed | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Candice A. Myers, Ph.D., Assistant Professor, Pennington Biomedical Research Center
Other Study IDs: 2017-060-PBRC; U54GM104940 (NIH)
Record Dates: First submitted 2018-01-26; First posted 2018-02-22 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Obesity; Psychological
Keywords: Food Insecurity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current pilot study will examine emergent hypotheses by investigating the role of psychological mechanisms in the relationship between food insecurity and obesity. This objective will be achieved via a cross-sectional, observational pilot study collecting quantitative and qualitative data.

DETAILED DESCRIPTION:
This pilot study will investigate an emergent risk factor for obesity: food insecurity, which is defined as the limited or uncertain availability of nutritionally adequate and safe foods. While paradoxically linked, numerous studies have shown a significant association between food insecurity and obesity. Moreover, recent narrative works have developed new, untested hypotheses linking food insecurity and obesity positing the causal role of psychological mechanisms. Given this, this mixed method pilot study will collect new psychological data in a sample of food secure and food insecure adults with and without obesity to examine the connections between food insecurity, body weight, and psychological constructs. The overarching objective of the study is to gather pilot data to identify potentially new intervention targets that will be used in future studies to more rigorously investigate the relationship between food insecurity and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years
* BMI ≥ 20.0 kg/m2
* Able to read and write using the English language
* Willing to provide written informed consent

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The target study sample will be 56 food secure and food insecure women and men aged 18 to 49 years with a BMI of 20.0 kg/m2 or greater.
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-28 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candice A Myers, Ph.D., Principal Investigator — Pennington Biomedicial Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

REFERENCES:
- [Derived] Myers CA, Beyl RA, Martin CK, Broyles ST, Katzmarzyk PT. Psychological mechanisms associated with food security status and BMI in adults: a mixed methods study. Public Health Nutr. 2020 Oct;23(14):2501-2511. doi: 10.1017/S1368980020000889. Epub 2020 Jun 29. PMID 32597739

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group: The study sample included a single group of 56 food secure and food insecure women and men aged 18 to 49 years with a BMI of 20.0 kg/m2 or greater.
Period: Overall Study
Arm/Group | Single Group
Started | 56
Completed | 56
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Group
Number analyzed (Participants) | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.25 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 27
  Caucasian or Asian American | 29
Region of Enrollment [Number; unit: participants]
  United States | 56

OUTCOME MEASURES:

1. Primary Outcome: Delay Discounting
Description: Assessed via the 27-Item Monetary Choice Questionnaire, which measures bias toward smaller, immediate rewards versus larger, delayed rewards. This questionnaire presents participants with a set of 27 choices between smaller, immediate monetary rewards and larger, delayed monetary rewards. Participants who discount the value of the delayed rewards more steeply are considered to be more impulsive. An estimate of a participant's discounting rate (k) is calculated from the pattern of choices. Values of k range from 0.00016 (ln transformation -8.74) to 0.25 (ln transformation -1.39), with higher values indicating a greater preference for smaller, immediate rewards over larger, delayed rewards. K tends to be skewed, so a natural log (ln) transformation is utilized to approximate a normal distribution for statistical analyses.
Time Frame: Through study completion, an average of 1 hour and 30 minutes at Study Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale (natural log)
Arm/Group | Single Group
Number analyzed (Participants) | 56
score on a scale (natural log) | -4.84 (2.07)

2. Secondary Outcome: Grit
Description: Assessed using the 8-item Short Grit Scale, which measures trait-level perseverance and passion for long-term goals. Scores range from 1 (not at all gritty) to 5 (extremely gritty).
Time Frame: Through study completion, an average of 1 hour and 30 minutes at Study Visit 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Group
Number analyzed (Participants) | 56
score on a scale | 3.68 (0.63)

ADVERSE EVENTS:
Time Frame: Through study completion, which was a single study visit with an average of 1 hour and 30 minutes.
Arm/Group | Single Group
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56
Other Adverse Events (participants affected / at risk) | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/94/NCT03441594/Prot_SAP_000.pdf